CLINICAL TRIAL: NCT00283361
Title: A Phase II,Randomized, Double-Blind, Flexible Dose Study of ZP120 I.V. Infusion as Add-On Therapy in Patients With Acute or Sub-Acute Decompensated Chronic Heart Failure NYHA Class III-IV Treated With Furosemide
Brief Title: ZP120 Add-on to Furosemide in Treatment of Acute or Sub-Acute Decompensated Heart Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Collaborators: Syneos Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-025
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2007-02-28 (Estimated); Status verified 2007-02

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure | interventions — ZP120; Blood Specimen Collection; Restraint, Physical

INTERVENTIONS:
Drug: ZP120
Procedure: I.v. catherization
Procedure: 6-minutes walk performance
Behavioral: Dyspnea severity assessment
Procedure: Blood sampling for laboratory tests
Procedure: ECG
Procedure: Physical examination

SUMMARY:
The main purpose of this study is to see if the experimental drug ZP120, when given with the approved drug furosemide to patients with acute or sub-acute heart failure, can reduce the amount of fluid in the patients' lungs and make breathing easier.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, age 18 years or more
2. A diagnosis of acute or subacute decompensated chronic heart failure, either ischemic or nonischemic, requiring hospitalization, and currently treated with furosemide, torsemide, or bumetadine, and other evidence based optimal treatment for heart failure. Patients must have the clinical diagnosis of CHF made at least 3 month prior to enrollment
3. Ambulatory
4. Objective signs of LVD corresponding to a LVEF < 45%, documented by any accepted method within the previous 12 months. If documentation is not available within the required time frame, LVEF must be assessed prior to enrollment
5. a) Worsening heart failure symptoms (current NYHA class III-IV). Patients must experience worsening of at least one of the symptoms described below at the time of entry into the study:

   Dyspnea Symptoms:
   * Dyspnea (labored or difficult breathing) at rest
   * Worsening dyspnea (labored or difficult breathing) on minimal exertion
   * Worsening orthopnea (difficult breathing except in the upright position)
   * Increased frequency of nocturnal dyspnea (awaken from sleep due to respiratory distress)

     b) Clinical evidence of volume overload such as weight gain over previous few days, peripheral edema, hepatic congestion with ascites, pulmonary congestion, or pleural effusion
6. Females of childbearing potential must have a negative pregnancy test at enrollment. A female is considered to be of childbearing potential unless she is post-menopausal (no menses for at least 12 consecutive months) or without a uterus and/or both ovaries
7. Ability to understand and willing to sign Informed Consent Form

Exclusion Criteria:

1. Incapable of taking the 6-minute walk test due to any condition unrelated to heart failure, e.g., muscular or skeletal disability
2. Valvular heart disease requiring surgical intervention (during the course of the study. Patients with heart failure due to or associated with uncorrected primary valvular disease, malfunctioning artificial heart valve, or uncorrected congenital heart disease)
3. History of or clinically significant evidence of any severe disease other than heart failure that preclude participation and complicate the evaluation of study results from the local laboratory:

   * Hepatic disease (AST, ALT, total bilirubin > 3 times Upper Limit of Normal (ULN), renal disease (S-Creatinine > 2.5 mg/dL),
   * Uncontrolled insulin-dependent diabetes mellitus with a history of frequent hypoglycemic episodes or frequent hospitalizations for hyperglycemia,
   * Cancer (excluding treated non-melanoma skin cancer)
4. Unstable angina, cardiogenic shock, or acute pulmonary edema requiring any of the following: Nitroprusside, intravenous nitroglycerin, nesiritide, intravenous inotrope, or need for endotracheal intubation and mechanical ventilation
5. Acute myocardial infarction and/or myocardial infarction within 30 days (prior to enrollment) as diagnosed by investigator's evaluation of clinical symptoms, ECG, and/or biochemical markers of cardiac injury
6. Cardiac arrest (patients with history of cardiac arrest within 12 months unless precipitated by an event such as an acute myocardial infarction, induction by catheter placement, severe transient electrolyte abnormality, by an electrophysiology procedure, or addressed by Automatic Implantable Cardioverter Defibrillator placement. Patients with increased risk of cardiac arrest, QTc > 450 msec, atrial ventricular block II or III, etc.)
7. Sustainable VT/VF within 30 days (> 15 seconds long; patients with enrollment ECG showing ventricular tachycardia or premature ventricular complexes associated with symptoms, or ventricular tachycardia of 6 beats)
8. Uncontrolled atrial fibrillation on enrollment ECG with a ventricular rate >120 bpm
9. Cardiac surgery within the last month or acutely required PCI (patients who have undergone a cardiac revascularization, valvular surgery, or biventricular resynchronization procedure within 30 days. Patients who have had ventricular reduction surgery or cardiac myoplasty and patients with mechanical ventricular assist device)
10. Systolic blood pressure < 90 mmHg and > 200 mmHg
11. Pulmonary embolism or DVT or history of pulmonary embolism or DVT within 6 months prior to enrollment
12. Severe obstructive or restrictive pulmonary disease, patients with primary pulmonary hypertension and heart failure secondary to pulmonary disease, and severe pulmonary infection
13. I.v. vasoactive treatment, e.g. vasodilators, positive inotropic agents, within 24 hours prior to enrollment (see details in Appendix E)
14. Participation in another study evaluating an experimental treatment within the last 30 days which potentially could bias the outcome of this study
15. Previous treatment with ZP120
16. Patients known to abuse or actively abusing alcohol or illicit drugs. Abuse of alcohol is defined as the usual daily intake of more than 100 grams of ethanol per day, or more than approximately six 12-ounce bottles of beer, one 750 mL bottle of wine, or 250 mL of 80 proof spirits
17. Inability or unwillingness to provide informed consent
18. BMI outside range of 20-50 kg/m2 (BMI equal to 20 and 50 kg/m2 is accepted)
19. Any other condition or therapy, which in the opinion of the Principal Investigator would make the patient unsuitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2006-01; Study Completion 2006-12

PRIMARY OUTCOMES:
Change in dyspnea severity

SECONDARY OUTCOMES:
Change in 6-minute walk test performance

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - LAC-USC Medical Center-Division of Cardiology, Los Angeles, California
  - VA Medical Center -WLA, Los Angeles, California
  - UCSD Medical Center, San Diego, California
  - San Francisco VA Medical Center, San Francisco, California
  - University of CO Health Sciences Center, Denver, Colorado
  - Health First Clinical Research Institute, Melbourne, Florida
  - Univ. of Miami Miller School of Medicine, Jackson Memorial Medical Center, Miami, Florida
  - Emory University Hospital/The Emory Clinic, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Community Hospital Anderson/Community Clinical Research Center, Anderson, Indiana
  - University of Iowa Heart Failure Treatment Program, Iowa City, Iowa
  - University of Maryland, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - The International Heart Institute, Missoula, Montana
  - Bryan LGH Heart Institute, Lincoln, Nebraska
  - University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Lancaster Heart Foundation, Lancaster, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Alamo Clinical Research Associates, San Antonio, Texas